CLINICAL TRIAL: NCT01960010
Title: A Phase 3, Multi-Center, Randomized, Double Masked, Placebo Controlled Clinical Study to Assess the Safety and Efficacy of 1% MIM-D3 Ophthalmic Solution in the Environment, and During Challenge in the Controlled Adverse Environmental (CAE) Model for the Treatment of Dry Eye
Brief Title: A Safety and Efficacy Study of MIM-D3 Ophthalmic Solution for the Treatment of Dry Eye
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mimetogen Pharmaceuticals USA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MIM-725
Record Dates: First submitted 2013-10-04; First posted 2013-10-10 (Estimated); Last update posted 2019-08-19 (Actual); Status verified 2019-08

CONDITIONS: Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1% MIM-D3 (Active Comparator): 1% MIM-D3 Ophthalmic Solution
  Interventions: Drug: MIM-D3 Ophthalmic Solution
- Vehicle (Placebo Comparator): Vehicle
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: MIM-D3 Ophthalmic Solution — 1% MIM-D3 dosed BID
  Other Names: Tavilermide Ophthalmic Solution
  Arms: 1% MIM-D3
Drug: Vehicle — Vehicle dosed BID
  Other Names: Placebo Ophthalmic Solution
  Arms: Vehicle

SUMMARY:
The purpose of this study is to assess the safety and efficacy of MIM-D3 Ophthalmic Solution compared with Placebo Ophthalmic Solution in treating the signs and symptoms of dry eye.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years of age
* Provided written informed consent
* Have a reported history of dry eye
* Have a history of use or desire to use eye drops for dry eye

Exclusion Criteria:

* Be diagnosed with an ongoing ocular infection (bacterial, viral, or fungal), or active ocular inflammation (e.g. follicular conjunctivitis) at Visit 1, or have been diagnosed with ocular rosacea, or any viral or bacterial disease of the cornea or conjunctiva, within the last 12 months
* Have any planned ocular and/or lid surgeries over the study period
* Have corrected visual acuity greater than or equal to +0.7 as assessed by Early Treatment of Diabetic Retinopathy Study (ETDRS) scale in both eyes at Visit 1
* Have an uncontrolled systemic disease
* Be a woman who is pregnant, nursing or planning a pregnancy
* Be a woman of childbearing potential who is not using an acceptable means of birth control; acceptable methods of contraception include: hormonal - oral, implantable, injectable, or transdermal contraceptives; mechanical - spermicide in conjunction with a barrier such as a diaphragm or condom; IUD; or surgical sterilization of partner. For non-sexually active females, abstinence may be regarded as an adequate method of birth control; however, if the subject becomes sexually active during the study, she must agree to use adequate birth control as defined above for the remainder of the study
* Have a known allergy and/or sensitivity to the test article or its components
* Have a condition or be in a situation which the investigator feels may put the subject at significant risk, may confound the study results, or may interfere significantly with the subject's participation in the study
* Be currently enrolled in an investigational drug or device study or have used an investigational drug or device within 45 days of Visit 1
* Be unable or unwilling to follow instructions, including participation in all study assessments and visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 403 (Actual)
Dates: Start 2013-10; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Corneal Fluorescein Staining | Day 29
Ocular Dryness | 28 Days
  Patient-derived, daily dryness symptoms for the 28 day time period will be be averaged to obtain a dryness score for the entire 28-day period. Average dryness scores over the 28-day treatment period will be compared between 1% MIM-D3 and placebo using t-tests.

SECONDARY OUTCOMES:
Total Ocular Fluorescein Staining | Day 29
Ocular Discomfort | 28 Days
  Patient-derived daily diary ocular discomfort symptoms for the 28 day time period will be averaged to obtain an ocular discomfort score for the entire 28-day period. Average ocular discomfort scores over the 28-day treatment period will be compared between 1% MIM-D3 and placebo using t-tests.

OTHER OUTCOMES:
Fluorescein staining (Ora CalibraTM Scale) | Day 15, 29 and 57
  Fluorescein Staining, (pre and post-CAESM; by individual region: central, superior, inferior, temporal, nasal, corneal sum, conjunctival sum, and total), by both grade and clearance of staining;
Lissamine green staining (Ora CalibraTM Scale,) | Day 15, 29 and 57
  Lissamine green staining (pre and post-CAESM; regions: central, superior, inferior, temporal, nasal, corneal sum, conjunctival sum, and total)
Subject diary individual symptoms | 28-day and 56-day treatment periods
Tear film break-up time | Day 15, 29 and 57
  Tear film break-up time (pre and post-CAESM);

CONTACTS AND LOCATIONS:
Overall Officials: Garth Cumberlidge, PhD, Study Director — Mimetogen Pharmaceuticals USA, Inc.
Locations (5):
- United States (5):
  - MIM-725 Investigational Site, Waterbury, Connecticut
  - MIM-725 Investigational Site, Lewiston, Maine
  - MIM-725 Investigational Site, Andover, Massachusetts
  - MIM-725 Investigational Site, Quincy, Massachusetts
  - MIM-725 Investigational Site, Memphis, Tennessee